CLINICAL TRIAL: NCT05704816
Title: The Effect of Different Types of Spinal Needles Used by First-year Anesthesia Residents on Procedural Success and Click Sensation: A Prospective, Observational Study
Brief Title: The Effect of Different Types of Spinal Needles on the Success of the Procedure
Status: Completed | Type: Observational
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Gamze Küçükosman, medical doctor, Zonguldak Bulent Ecevit University
Other Study IDs: 2018/20
Record Dates: First submitted 2022-10-03; First posted 2023-01-30 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Spinal Needle Diameter and Design, Click Feeling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Quincke (Q)-25 Gauge
  Interventions: Other: Spinal anesthesia application
- Quincke (Q)-26Gauge
  Interventions: Other: Spinal anesthesia application
- Quincke (Q)-27 Gauge
  Interventions: Other: Spinal anesthesia application
- Pencil-point (P)-25Gauge
  Interventions: Other: Spinal anesthesia application
- Pencil-point (P)-26Gauge
  Interventions: Other: Spinal anesthesia application
- Pencil-point (P)-27Gauge
  Interventions: Other: Spinal anesthesia application

INTERVENTIONS:
Other: Spinal anesthesia application — The success of the needles with different tip designs and thicknesses used in spinal anesthesia application

SUMMARY:
The effects of spinal needles with different tip designs on the success of the application and the number of attempts required to get the spinal click feeling.

ELIGIBILITY:
Inclusion Criteria:

* Elective lower abdomen/extremity surgery planned,
* American Society of Anesthesiologists (ASA) I-II risk group,
* without bleeding diathesis
* patients with written consent

Exclusion Criteria:

* Patients for whom spinal anesthesia is contraindicated,
* morbidly obese,
* pregnant
* Patients with a history of allergic reactions to the drugs used in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 213
Sampling Method: Non-Probability Sample
Enrollment: 213 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
The Effect of Different Types of Spinal Needles Used by First-year Anesthesia Residents on Procedural Success and Click Sensation: A Prospective, Observational Study | Spinal anesthesia procedure time
  Clicking feeling: Considering that the click feeling due to dural puncture is taken, in which attempt (1, 2, and ≥3) the needle's guide was removed and the cerebrospinal fluid (CSF) arrival occurred Procedural success: Time until CSF is seen (<1.9sec, ≥2sec)
The Effect of Different Types of Spinal Needles Used by First-year Anesthesia Residents on Procedural Success and Click Sensation: A Prospective, Observational Study | Spinal anesthesia procedure time
  Procedural success: Time until CSF is seen (<1.9sec, ≥2sec)

SECONDARY OUTCOMES:
The Effect of Different Types of Spinal Needles Used by First-year Anesthesia Residents on Procedural Success and Click Sensation: A Prospective, Observational Study | Spinal anesthesia procedure time
  First-year anesthesia assistants get a click feeling with needles with different tip designs and diameters

CONTACTS AND LOCATIONS:
Locations (1):
- Gamze Küçükosman, Zonguldak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No